CLINICAL TRIAL: NCT04019821
Title: Effects of Super-Bolus on Postprandial Glycemia After High Glycemic Index Meal in Children With Type 1 Diabetes Mellitus- Randomized Study
Brief Title: Super-Bolus: Effects on Postprandial Glycemia After High Glycemic Index Meal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SuperBolus
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: super bolus; diabetes type 1; insulin bolus; high glycemic index meal; prandial insulin requirement; postprandial glycemia; insulin pump therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — insulin glulisine; Insulin Aspart; Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Normal Bolus (Active Comparator): Pre-breakfast insulin will be given as a Normal Bolus 15 minutes before the high-glycemic index meal (cornflakes and milk). The Normal Bolus will be calculated based on individual insulin-to-carbohydrate ratio (ICR).
  Interventions: Drug: Insulin Glulisine; Drug: Insulin Aspart; Drug: Insulin Lispro
- Super Bolus (Experimental): Pre-breakfast insulin will be given as a Super Bolus 15 minutes before the high-glycemic index meal (cornflakes and milk). The Super Bolus will be calculated based on individual ICR increased to 150% and basal insulin will be suspended for 2 hours at the same time.
  Interventions: Drug: Insulin Glulisine; Drug: Insulin Aspart; Drug: Insulin Lispro

INTERVENTIONS:
Drug: Insulin Glulisine — A type of bolus insulin will be insulin glulisine if participant used insulin glulisine before entering the trial.
  Other Names: Apidra
Drug: Insulin Aspart — A type of bolus insulin will be insulin aspart if participant used insulin aspart before entering the trial.
  Other Names: NovoRapid
Drug: Insulin Lispro — A type of bolus insulin will be insulin lispro if participant used insulin lispro before entering the trial.
  Other Names: Humalog, Liprolog

SUMMARY:
The aim of this study is to determine whether Super-Bolus is more effective in postprandial glycemic control than Normal-Bolus after the high glycemic index (H-GI) meal in children with type 1 diabetes (T1DM) treated with insulin pump (continuous subcutaneous insulin infusion, CSII).

ELIGIBILITY:
Inclusion Criteria:

* duration of type 1 diabetes longer than 12months,
* insulin pump therapy longer than 3 months,
* written informed consent to participate in the study signed by parents (and patient older than 16 years).

Exclusion Criteria:

* celiac disease,
* diabetes related complications (e.g. nephropathy),
* BMI at or above the 95th percentile and at or below 3rd percentiles for children and teenagers of the same age and sex,
* withdrawal of consent to participate in the study,
* comorbid conditions and treatment which could significantly affect glycemic values in the researchers' opinion.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Postprandial Glycemia | 90 minutes after the prandial bolus
  Postprandial blood glucose excursion measured by self monitoring of blood glucose (SMBG)

SECONDARY OUTCOMES:
Hypoglycemia Episodes | 3-hours after the prandial bolus
  Hypoglycemia defined as a plasma glucose concentration below or equal 70mg/dl with or without symptoms
Glucose Area Under the Curve (AUC) | 3-hours after the prandial bolus
  Measurements based on Continuous Glucose Monitoring System (CGMS)
Mean amplitude of glycaemic excursion (MAGE) | 3-hours after the prandial bolus
  MAGE will be defined as a standard deviation of blood glucose (SDBG) obtained from all blood glucose concentrations
Capillary blood glucose level 30,60,120,150,180 min after administration of the prandial bolus | 3-hours after the prandial bolus
  measured by SMBG
Glycemic rise (GR) | 3-hours after the prandial bolus
  a difference between baseline and the maximum glucose value based on CGMS
Peak glucose level (PG) | 3-hours after the prandial bolus
  the maximum value of glycemia during 3 hours of postmeal time based on CGMS
Time to glucose peak | 3-hours after the prandial bolus
  based on CGMS
Time in postprandial glucose range between 70 to 180 mg/dl (4.0-10.0 mmol/L) | 3-hours after the prandial bolus
  based on CGMS

CONTACTS AND LOCATIONS:
Overall Officials: Agnieszka Szypowska, Prof., Study Chair — Department of Pediatrics, Medical University of Warsaw
Locations (1):
- Department of Pediatric Diabetology and Pediatrics, Pediatric Teaching Clinical Hospital, Warsaw, Poland

REFERENCES:
- [Derived] Kowalczyk-Korcz E, Dyminska M, Szypowska A. Super Bolus-A Remedy for a High Glycemic Index Meal in Children with Type 1 Diabetes on Insulin Pump Therapy?-A Randomized, Double-Blind, Controlled Trial. Nutrients. 2024 Jan 16;16(2):263. doi: 10.3390/nu16020263. PMID 38257156
- [Derived] Kowalczyk E, Dzygalo K, Szypowska A. Super Bolus: a remedy for a high glycemic index meal in children with type 1 diabetes on insulin pump therapy?-study protocol for a randomized controlled trial. Trials. 2022 Mar 29;23(1):240. doi: 10.1186/s13063-022-06173-4. PMID 35351180